CLINICAL TRIAL: NCT02866019
Title: A Phase III, Multicenter, Open-label Study to Evaluate the Esophageal Stenosis Inhibition Effects and Safety of CLS2702C/CLS2702D After Endoscopic Submucosal Dissection (ESD) in Patients With Superficial Esophageal Cancer
Brief Title: Human (Autologous) Oral Mucosal Cell Sheet Transplantation After ESD in Patients With Superficial Esophageal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CellSeed Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLS2702-ESO-01
Record Dates: First submitted 2016-08-05; First posted 2016-08-15 (Estimated); Last update posted 2019-03-07 (Actual); Status verified 2019-02

CONDITIONS: Superficial Esophageal Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CLS2702C/CLS2702D (Experimental)
  Interventions: Device: CLS2702C/CLS2702D

INTERVENTIONS:
Device: CLS2702C/CLS2702D — CLS2702C (cell sheet) will be transplanted to the wound site using CLS2702D (transplantation device) (screening period, 1 month [4 weeks]; cell sheet culture period, 0.5 month [16 days]; transplantation period, assessment/follow-up period, 6 months [24 weeks])
  Other Names: Human (autologous) oral mucosal cell sheet; Transplantation device

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of esophageal epithelial regenerative treatment by the transplantation of the product, CLS2702C, to the esophageal wound site after extensive ESD for superficial esophageal cancer.

DETAILED DESCRIPTION:
This study is a multicenter, single-arm, open-label study of CLS2702C/D in patients who plan to undergo ESD for superficial esophageal cancer.

In this study, the efficacy and safety of CLS2702C (cell sheet) transplanted (applied) to the wound site after ESD using CLS2702D (transplantation device) will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who plan to undergo ESD for the treatment of superficial esophageal cancer
2. Patients aged ≥20 years at the time of consent
3. Patients with no clinical metastasis (cN0M0) by cervical to abdominal CT
4. Patients with an endoscopically diagnosed depth of wall invasion remaining in the epithelium (EP) or lamina propria mucosae (LPM)
5. Patients with ≥3/4 of circumference and a length of <8 cm
6. If the patient has multiple lesions, the circumference of all minor lesions other than the one lesion with the largest circumference (major lesion) must be <1/2, and the distance between the minor lesions and the major lesion must be 5 cm or more on the major axis.
7. Patients with squamous cell carcinoma (including high-grade intraepithelial neoplasia) as confirmed by biopsy
8. Patients whose lesion is confirmed to be localized in the thoracic esophagus (lesions in the cervical esophagus or abdominal esophagus will be excluded). The location of the lesion will be determined by endoscopy.
9. Patients who have not received pretreatment for esophageal cancer. Treatment by ESD for superficial esophageal cancer for which the depth of wall invasion has been assessed to remain in the epithelium (EP) or lamina propria mucosae (LPM) is not included in the definition of pretreatment. However, patients who have a scar due to previous ESD in the major or minor lesions will be excluded from the study.
10. Patients with an ECOG Performance Status (PS) of 0 or 1
11. Patients in whom a commonly used endoscope with a tip diameter of 8.9 mm can pass
12. Patients with a dysphagia score of 0
13. Patients whose laboratory values within 28 days before enrolment meet all of the following criteria:

    * White blood cell count: ≥4,000/µL
    * Platelet count: ≥100,000/µL
    * AST: ≤100 IU/L
    * ALT: ≤100 IU/L
    * Total bilirubin: ≤2.0 mg/dL
    * Serum creatinine: ≤2.0 mg/dL
14. Patients who have received sufficient explanation about the study and provided written voluntary consent

Exclusion Criteria:

1. Patients with cardiac disease (myocardial infarction, unstable angina, and heart failure), renal disease (nephrotic syndrome and kidney failure), or poorly controlled diabetes mellitus
2. Patients who have an active (within 1 year) malignancy other than esophageal cancer
3. Patients with active bacterial, fungal, or viral infection
4. Patients who are being treated with a corticosteroid
5. Patients with positive HBs antigen, positive HCV antibody, positive HIV antibody, positive HTLV antibody, or positive Treponema pallidum (tested at screening). For patients with positive HBc/HBs antibody, HBV-DNA test will be performed (if the result is negative, the patient will be allowed to enter the study).
6. Patients with a mental disorder that is difficult to control
7. Pregnant women, lactating women, and potentially pregnant women

   * Lactating women may be enrolled in the study if they discontinue lactation during the period from trans-plantation to confirmed wound healing.
   * Women of childbearing potential must agree to use the following birth control methods or completely ab-stain from sexual intercourse during the period from consent to participate in the study to the end of study participation.

     * Principal birth control methods: oral contraceptives, intrauterine contraceptive devices including intrauterine luteal hormone-releasing systems, tubal occlusion, and vasectomized partner
     * Supportive birth control methods: condoms and diaphragms
   * The use of principal birth control methods is essential. Supportive birth control methods should not be used alone and must be used together with the principal birth control methods. For oral contraceptives, changes in the birth control methods or other strategies should be considered because it is known that their effect is reduced if they are missed or concomitantly taken with certain types of drugs or dietary supplements.
8. Patients who have participated in another clinical study within 6 months, those who are participating in another clinical study, and those who plan to participate in another clinical study during participation in Study CLS2702-ESO-01
9. Patients from whom tissues cannot be collected due to a disease (e.g., stomatitis, erosion, mass, and blister) in the oral mucosa at the tissue collection site
10. Patients with a history of hypersensitivity to antibiotic preparations (ampicillin sodium, sulbactam sodium, streptomycin sulfate, gentamicin sulfate, or amphotericin B) or who have taken drugs that may affect the study (within 28 days before enrolment)
11. Patients who have undergone radiotherapy in the cervical to upper abdominal region, or surgery for head and neck cancer that may affect the assessment of ESD or stenotic symptoms
12. Patients whose swallowing function has been markedly reduced or completely lost due to a sequela of cerebral infarction or other reasons
13. Patients with porcine or latex allergy
14. Patients who, in the opinion of the treating physician, are not eligible for the study due to reasons other than those described above

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Proportion of participants without stenosis until 8 weeks after endoscopic submucosal dissection (ESD) | Up to 8 weeks after ESD

SECONDARY OUTCOMES:
Time to wound healing | Up to 24 weeks after ESD
  Wound healing is defined as re-epithelized state with no white coat, erosion, or ulcer in the process of healing. The time to wound healing will be assessed endoscopically.
Number of esophageal balloon dilatations (investigated until wound healing is confirmed) | Up to 24 weeks
  Number of esophageal balloon dilatations will be counted.
Number of participants reporting one or more adverse events and product deficiencies | From day -16 to 24 weeks
  An adverse event is defined as any untoward medical occurrence in a subject who has used the product or received the study treatment, regardless of the causal relationship with the product.
  An adverse event can therefore be any untoward and unintended sign (including abnormal laboratory finding), symptom, or disease (new disease or worsening of an existing disease) temporally associated with the use of the product or implementation of the study treatment.
Quality of Life (QOL) measured with the EORTC QLQ-C30 | Up to 4 weeks
  The European Organization for Research and Treatment of Cancer QLQ-C30 is a quality-of-life instrument for use in international clinical trials in oncology. The QLQ-C30 incorporates nine multi-item scales: five functional scales (physical, role, cognitive, emotional, and social); three symptom scales (fatigue, pain, and nausea and vomiting); and a global health and quality-of-life scale.
QOL assessed by the EORTC QLQ-OG 25 | Up to 24 weeks
  EORTC QLQ-OG25 questionnaire is a quality-of-life instrument for use in patients with esophagogastric cancers. The QLQ-OG25 has six scales, dysphagia, eating restrictions, reflux, odynophagia, pain and anxiety.

CONTACTS AND LOCATIONS:
Locations (3):
- Japan (3):
  - National Cancer Center Hospital East, Kashiwa-shi, Chiba
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - Tokyo Women's Medical University Hospital, Shinjuku-ku, Tokyo